CLINICAL TRIAL: NCT01594385
Title: Seprafilm in Open Abdomens: a Prospective Evaluation of Wound and Adhesion Characteristics in Trauma Damage Control (OASIT)
Brief Title: Seprafilm in Open Abdomens: a Study of Wound and Adhesion Characteristics in Trauma Damage Control Patients
Acronym: OASIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stan Stawicki (Other)
Responsible Party: Sponsor-Investigator, Stan Stawicki, Associate Professor of Surgery, St. Luke's Hospital and Health Network, Pennsylvania
Organization: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009H0311
Record Dates: First submitted 2012-01-05; First posted 2012-05-09 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Open Abdomen; Abdominal Adhesions; Trauma; Wounds and Injury
Keywords: Open Abdomen; Damage Control; Trauma; Wound healing; Gun shot wounds; Stab wounds; Automobile accidents; Wounds and Injury
MeSH Terms: conditions — Wounds and Injuries; Wounds, Stab | interventions — Seprafilm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seprafilm (Other): The treatment group will receive Seprafilm while the control group will not receive Seprafilm. Allocation of patients will be in 1:1 ratio.
  Interventions: Biological: Seprafilm
- No Seprafilm (No Intervention): This group will be treated according to the current standard of care. No seprafilm will be applied in this subset of patients.

INTERVENTIONS:
Biological: Seprafilm — Two sheets of the Seprafilm material will be applied at each reoperation. Each sheet will be cut into 1x1 inch squares and applied to the following anatomic areas:
  * Two Seprafilm pieces between the liver and the anterior abdominal wall
  * Four pieces over the exposed bowel surfaces anteriorly
  * Two slightly staggered pieces of Seprafilm in each colic gutter
  * Two pieces in the pelvic area.
  * If any of the above areas involve an anastomosis or bowel repair, then the Seprafilm should be placed at least 1 inch away from the anastomosis and/or bowel repair.
  Arms: Seprafilm

SUMMARY:
The goal of this study is to test the effects of Seprafilm adhesion barrier on patients who are undergoing open abdomen damage control management for traumatic injuries when compared to no adhesion barrier use. Specifically, the researchers wish to study the effects of Seprafilm adhesion barrier on:

* the number and intensity of adhesions,
* whether there is any difference between treatment groups (Seprafilm vs. no Seprafilm) who go on to successful definitive abdominal closure,
* rate of occurrence of secondary complications (such as abscesses) associated with short- and long-term beneficial effects of reducing adhesion formation,and
* whether there is any difference between treatment groups regarding patient functional recovery.

DETAILED DESCRIPTION:
Data to be analyzed includes:

Age, gender, traumatic injuries, trauma alert level, procedure information, length of hospital stay, length of ICU stay, interval between admission and initial operation, interval between operations, whether operation took place during the day or night, duration of operation in minutes, number of surgeons present during the operation, description of the initial operation, justification for using damage control approach, complications noted, injuries missed or delayed in diagnosis, Acute Physiology and Chronic Health Evaluation II (APACHE II) calculations at various time points, Simplified Acute Physiology Score (SAPS II) calculations at various time points, Glasgow Coma Score (GCS) calculations at various time points, changes in GCS at over time, Injury Severity Score (ISS) at various time points, Abbreviated Injury Scale (AIS) at various time points, Penetrating Abdominal Trauma Index score (if applicable) at various time points, complete blood count (CBC) results at various time points, blood chemistry results at various time points, blood gas results at various time points, subject randomization information, number of operations, adhesion scores (Zuhlke and Yaacobi) for each operative procedure, contamination score for each operative procedure, diagnosis and description of sub-procedures for each operative procedure, wound characteristics from the start and end of all operative procedures (e.g. length and width of the fascia and skin), type of abdominal coverage or closure, discharge destination (e.g. home, short term rehabilitation facility, etc.), Functional Outcome Measure score, Glasgow Outcome Score (GOS) at various time points, number and interval of post discharge follow-up visits, wound characteristics since discharge at several time points and complications/complaints noted since discharge at several time points.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients undergoing DC/OA management for traumatic injury
* Age 18+
* Life expectancy longer than 48 hours

Exclusion Criteria:

* Prisoners
* Pregnant patients
* Younger than 18 years of age

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw P Stawicki, MD, Principal Investigator — Ohio State University
Locations (5):
- United States (5):
  - Cooper University Hospital, Camden, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Currently, the only available data is de-identified dataset without any linkages to the original data. Data storage currently past record-keeping requirements. Study was permanently closed in June 2014.

REFERENCES:
- [Result] Stawicki SP, Green JM, Martin ND, Green RH, Cipolla J, Seamon MJ, Eiferman DS, Evans DC, Hazelton JP, Cook CH, Steinberg SM; OPUS 12 Foundation, Inc, Multi-Center Trials Group & OASIT Investigators. Results of a prospective, randomized, controlled study of the use of carboxymethylcellulose sodium hyaluronate adhesion barrier in trauma open abdomens. Surgery. 2014 Aug;156(2):419-30. doi: 10.1016/j.surg.2014.03.007. Epub 2014 Mar 15. PMID 24962185

RESULTS

PARTICIPANT FLOW:
Groups:
- Seprafilm Group: Patient who randomized to this group received seprafilm at the end of each consecutive operation; Seprafilm from each previous operation was washed out at the beginning of each subsequent re-operation.
- No Seprafilm Group: Patients randomized to this group received no Seprafilm; Abdominal washout at the beginning of each procedure was performed in a fashion identical that in the Seprafilm Group.
Period: Overall Study
Arm/Group | Seprafilm Group | No Seprafilm Group
Started | 17 | 13
Completed | 17 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Seprafilm: The treatment group will receive Seprafilm while the control group will not receive Seprafilm. Allocation of patients will be in approximately 1:1 ratio.
  Seprafilm: Two sheets of the Seprafilm material will be applied at each reoperation. Each sheet will be cut into 1x1 inch squares and applied to the following anatomic areas:
  * Two Seprafilm pieces between the liver and the anterior abdominal wall
  * Four pieces over the exposed bowel surfaces anteriorly
  * Two slightly staggered pieces of Seprafilm in each colic gutter
  * Two pieces in the pelvic area.
  * If any of the above areas involve an anastomosis or bowel repair, then the Seprafilm should be placed at least 1 inch away from the anastomosis and/or bowel repair.
- No Seprafilm: Patients in this group will not receive Seprafilm during re-operations. Otherwise, their surgical management will be identical to the Seprafilm Group.
- Total: Total of all reporting groups
Arm/Group | Seprafilm | No Seprafilm | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (16.7) | 40.2 (16.3) | 40.3 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Adhesion Characteristics
Description: Zuhlke adhesion score (1 - minimum to 4 - maximum)
  1. = filmy adhesions, easy to separate by blunt dissection
  2. = stronger adhesions; blunt dissection possible, partly sharp dissection necessary; beginning of vascularization
  3. = strong adhesions; lysis possible by sharp dissection only; clear vascularization
  4. = very strong adhesions; lysis possible by sharp dissection only; organs strongly attached with severe adhesions; damage to organs hardly preventable
Time Frame: Up to 1 year
Measure: Mean (Standard Error); unit: Scores on a scale
Units Other Than Participants: Zuhlke Adhesion Score
Groups:
- Seprafilm: Operation Number Zuhlke scores (mean / standard error) Operation #1 1.06 / 0.24 Operation #2 1.13 / 0.34 Operation #3 1.54 / 0.69 Operation #4 1.39 / 0.49 Operation #5 1.21 / 0.39 Operation #6 1.50 / 0.77 Operation #7 1.38 / 0.25
- No Seprafilm: Operation Number Zuhlke scores (mean / standard error) Operation #1 1.08 / 0.28 Operation #2 1.08 / 0.28 Operation #3 1.19 / 0.32 Operation #4 1.63 / 0.58 Operation #5 2.33 / 0.82 Operation #6 2.92 / 0.83 Operation #7 2.84 / 0.23
Arm/Group | Seprafilm | No Seprafilm
Number analyzed (Participants) | 17 | 13
Number analyzed (Zuhlke Adhesion Score) | 62 | 58
Scores on a scale
  Operation 1 | 1.06 (0.24) | 1.08 (0.28)
  Operation 2 | 1.13 (0.34) | 1.08 (0.28)
  Operation 3 | 1.54 (0.69) | 1.19 (0.32)
  Operation 4 | 1.39 (0.49) | 1.63 (0.58)
  Operation 5 | 1.21 (0.39) | 2.33 (0.82)
  Operation 6 | 1.50 (0.77) | 2.92 (0.83)
  Operation 7+ | 1.38 (0.25) | 2.84 (0.23)

2. Secondary Outcome: Wound Healing Characteristics
Description: There will not be a fixed duration of outpatient follow-up (fixed follow-up in trauma patients is not practical due to the unpredictable nature of trauma population), an average (mean) follow-up will be determined for the entire cohort of patients for the purposes of the study, up to a maximum of 1 year (if available) following hospital discharge.
Time Frame: Participants will be followed until their open abdomen is closed. Depending on the nature and severity of the wound, this period may last as long as 1 year after the patient has been discharged.
Population: Wound areas for Seprafilm and "No Seprafilm" groups were obtained serially, by measuring each wound horizontally and vertically and multiplying measurements (in centimeters) to determine the estimated area in cm squared.
Measure: Mean (Standard Deviation); unit: Square Centimeters (cm2)
Groups:
- Wound Sizes: Seprafilm: Wound size characteristics (estimated area = "Width x Length" in centimeters squared) for patients who received Seprafilm
- Wound Sizes: No Seprafilm: Wound size characteristics (estimated area = "Width x Length" in centimeters squared) for patients who did not receive Seprafilm
Arm/Group | Wound Sizes: Seprafilm | Wound Sizes: No Seprafilm
Number analyzed (Participants) | 17 | 13
Square Centimeters (cm2)
  Composite wound size (cm2): Time 0 | 419 (238) | 393 (225)
  Composite wound size (cm2): Week 02 | 282 (224) | 322 (231)
  Composite wound size (cm2): Week 04 | 223 (278) | 218 (199)
  Composite wound size (cm2): Week 08 | 76 (70) | 210 (176)
  Composite wound size (cm2): Week 12 | 35 (5) | 116 (28)
  Composite wound size (cm2): Week 24 | 66 (30) | 148 (106)
  Composite wound size (cm2): Week 32 | 64 (55) | 59 (36)

3. Other Pre Specified Outcome: Patient Mortality
Description: Assessment of patient mortality at 28 days, with subsequent determination of survival (i.e., patient status at last known follow-up)
Time Frame: 28 days & end of follow-up
Population: Note: Both mortalities in the Seprafilm group involved withdrawal of care as per previously stated patient wishes.
Measure: Number; unit: Mortalities
Groups:
- Seprafilm: The treatment group will receive Seprafilm.
Arm/Group | Seprafilm | No Seprafilm
Number analyzed (Participants) | 17 | 13
Mortalities | 2 | 1

4. Other Pre Specified Outcome: Enterocutaneous and Other Fistula
Description: Determination of enterocutaneous/other fistula among study patients during the hospitalization and the follow-up interval
Time Frame: Up to 1 year post-injury
Measure: Number; unit: Total events
Arm/Group | Seprafilm | No Seprafilm
Number analyzed (Participants) | 17 | 13
Total events | 3 | 6

5. Other Pre Specified Outcome: Ventral Hernia
Description: Determination of ventral hernia presence during follow-up visits
Time Frame: Up to 1 year follow-up
Measure: Number; unit: Hernia
Arm/Group | Seprafilm | No Seprafilm
Number analyzed (Participants) | 17 | 13
Hernia | 1 | 0

6. Other Pre Specified Outcome: Infection / Abscess / Sepsis
Description: Assessment of any infection, abscess, or sepsis during the initial and the follow-up periods
Time Frame: Up to 1 year
Measure: Number; unit: Total events
Arm/Group | Seprafilm | No Seprafilm
Number analyzed (Participants) | 17 | 13
Total events | 4 | 3

7. Other Pre Specified Outcome: Bowel Obstruction
Description: Determination of bowel obstruction during the entire available study follow-up period
Time Frame: Up to 1 year follow-up
Measure: Number; unit: Bowel obstruction
Arm/Group | Seprafilm | No Seprafilm
Number analyzed (Participants) | 17 | 13
Bowel obstruction | 0 | 1

8. Other Pre Specified Outcome: Patient Functional Outcomes
Description: Assessment of Glasgow Outcome Scale (GOS) and the Functional Outcome Measures (FOM) during the available follow-up period.
  FOM Source: [1] Ohio Dept of Public Safety. Ohio Trauma Registry Data Dictionary. Columbus: 2004.
  FOM Scale range: 1 (worst) to 4 (best); GOS Scale: 1 (worst) to 5 (best)
  FOM Feeding Subscale
  1. Fully dependent
  2. Partially dependent
  3. Independent w/device
  4. Fully independent
  FOM Locomotion Subscale
  1. Fully dependent
  2. Partially dependent
  3. Independent w/device
  4. Fully independent
  FOM Expression/Communication Subscale
  1. Fully dependent
  2. Partially dependent
  3. Independent w/device
  4. Fully independent
  Glasgow Outcome Scale:
  1. Death
  2. Persistent vegetative state: Minimal responsiveness
  3. Severe disability: Conscious but disabled; dependent on others for daily support
  4. Moderate disability: Disabled but independent; can work in sheltered setting
  5. Good recovery: Resumption of normal life despite minor deficits
Time Frame: Up to 1 year follow-up
Population: Please see Outcome Measure Description [above] for exact measure(s) utilized, including measurement scale(s).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seprafilm | No Seprafilm
Number analyzed (Participants) | 17 | 13
units on a scale
  Self-Feeding Score | 2.93 (1.44) | 3.25 (1.14)
  Locomotion Score | 2.6 (1.24) | 2.25 (0.87)
  Expression / Communication | 3.47 (1.13) | 3.45 (1.21)
  Glasgow Outcome Score | 4.07 (0.80) | 3.40 (0.97)

9. Other Pre Specified Outcome: Would Complication
Description: Tracking of wound infection, dehiscence, hernia, or any other would-related complication of complaint
Time Frame: Up to 1 year follow-up period
Measure: Number; unit: Wound complication
Arm/Group | Seprafilm | No Seprafilm
Number analyzed (Participants) | 17 | 13
Wound complication | 5 | 3

ADVERSE EVENTS:
Time Frame: Daily assessments for adverse events (AE) were performed during the initial hospitalization phase for each patient; Additional AE screening was done during outpatient visits; AE data were collected during up to 1 year voluntary follow-up.
Arm/Group | Seprafilm Group | No Seprafilm Group
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/13
Other Adverse Events (participants affected / at risk) | 5/17 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seprafilm Group (N=17) | No Seprafilm Group (N=13)
Mortality (Surgical and medical procedures) | 2 | 1 — Two patients (2/17) in the Seprafilm group experienced 28-day mortality; One patient (1/13) in No Seprafilm group experienced 28-day mortality; Mortality was attributed to high injury severity and physiologic acuity; Not associated with the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Seprafilm Group (N=17) | No Seprafilm Group (N=13)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5 — 5/17 patients in Seprafilm group developed respiratory failure; 5/13 in No Seprafilm group developed respiratory failure; All instances of respiratory failure were related to injury severity / physiologic acuity; Not related to study conduct

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No